CLINICAL TRIAL: NCT03804008
Title: The Efficacy of Fundamental Advice and a Heel Cup Versus Fundamental Advice and a Heel Cup Plus eXercise Versus Fundamental Advice and a Heel Cup Plus Exercise and a Corticosteroid Injection in Individuals With Plantar Fasciopathy
Brief Title: Advice vs Advice + Exercise vs Advice + Exercise + Injection for Individuals With Plantar Fasciopathy
Acronym: FIX-Heel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Henrik Riel, PhD student, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20180066
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Plantar Fasciopathy

STUDY DESIGN:
Masking Description: Analyses will be carried out by a blinded data analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fundamental advice and a heel cup (Active Comparator)
  Interventions: Other: Fundamental advice and a silicone heel cup
- Fundamental advice and a heel cup plus exercise (Active Comparator)
  Interventions: Other: Heavy-slow resistance training; Other: Fundamental advice and a silicone heel cup
- Fundamental advice and a heel cup plus exercise and injection (Active Comparator)
  Interventions: Drug: Ultrasound-guided corticosteroid injection; Other: Heavy-slow resistance training; Other: Fundamental advice and a silicone heel cup

INTERVENTIONS:
Drug: Ultrasound-guided corticosteroid injection — A 21-gauge, 40 mm needle is connected to a 2.5 cm3 syringe filled with 1 ml Triamcinolonhexacetonid 20mg/ml + 1 ml Lidocain 10 mg7ml. The skin is cleansed with Chlorhexidine alcohol 0.5 %. The needle is inserted with a medial approach under ultrasound-guidance aligned to the long axis of the ultrasound transducer. The injection is placed anterior to the plantar fascia insertion on the calcaneal bone in the region of maximal fascia thickness. Participants are asked to start performing the exercise as soon as they feel ready but not before 24 hours after the injection. Furthermore, they are asked not to progress the method used to achieve 8RM when they start to do the exercise after the injection until Week 3 of the exercise programme. If standing on both feet was sufficient to achieve 8RM at baseline, the participant must not perform the exercise single-legged or to wear a backpack with weights after the injection regardless of any pain reduction afforded by the injection.
  Arms: Fundamental advice and a heel cup plus exercise and injection
Other: Heavy-slow resistance training — Participants will be asked to complete a heel raise standing with the forefoot on a step. The toes are maximally dorsi flexed by placing a towel underneath them. The participant is instructed to perform a heel raise to maximal plantar flexion in the ankle joint and afterwards to lower the heel to maximal dorsiflexion. Supporting oneself for balance by placing the hands on a wall or a rail is allowed. Participants are instructed in performing the exercise with a load as heavy as possible but no higher than 8RM and for as many sets as possible every other day.
  Arms: Fundamental advice and a heel cup plus exercise; Fundamental advice and a heel cup plus exercise and injection
Other: Fundamental advice and a silicone heel cup — Participants receive brief information about pathology, risk factors and advice on how to decrease activities that lead to symptom flares and slowly increase their activity level based on their symptoms. They also receive a leaflet that includes the same information as the research assistants will deliver orally after inclusion and a silicone heel cup.

SUMMARY:
The purpose of this trial is to investigate the efficacy of fundamental patient advice and a heel cup versus fundamental patient advice and a heel cup plus heavy-slow resistance training versus fundamental patient advice and a heel cup plus heavy-slow resistance training and an ultrasound-guided corticosteroid injection in improving the Foot Health Status Questionnaire pain domain score in individuals with plantar fasciopathy after 12 weeks.

DETAILED DESCRIPTION:
This trial will be designed as a randomised, data analyst-blinded, superiority trial, with a 3-group parallel design to be conducted in Aalborg, Denmark. Reporting of the trial will follow CONSORT guidelines and TIDieR for intervention description. Reporting of the protocol will follow the SPIRIT statement. The planning of the trial is done in accordance with the PREPARE Trial guide.

Participants will be stratified by sex and block randomised in block sizes of 3 to 12 (1:1:1) into 3 parallel groups of 60 participants using a random number generator on www.sealedenvelope.com. The block sizes will be random and concealed to the research assistants responsible of including participants. Group allocation will be coded, and the data analyst will be blinded to this code until after the analyses have been performed.

The investigators will only conclude superiority of one intervention over the other if the intention-to-treat analysis leads to mean between-group differences of the Foot Health Status Questionnaire pain domain ≥14 points (minimally important difference) and P-values <0.05 at the primary endpoint (12 weeks) after adjustment for the baseline value.

ELIGIBILITY:
Inclusion Criteria:

* history of inferior heel pain for at least three months before enrolment
* pain on palpation of the medial calcaneal tubercle or the proximal plantar fascia
* thickness of the plantar fascia of 4.0 mm or greater as measured by ultrasonography
* mean heel pain of ≥30 mm on a 100 mm VAS during the previous week

Exclusion Criteria:

* below 18 years of age
* diabetes
* history of inflammatory systemic diseases
* pregnancy or breastfeeding
* corticosteroid injection for plantar fasciopathy within the previous six months
* pain or stiffness in the 1st metatarsophalangeal joint to an extent where the exercises cannot be performed
* known hypersensitivity to corticosteroids or local anaesthetics
* skin or soft tissue infection near the injection site
* received treatment by a healthcare professional for plantar fasciopathy within the previous 12 weeks
* made any substantial changes to usual self-care of the condition in the last 4 weeks (e.g. started using insoles, started performing stretching, made a substantial decrease in physical activity level)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Change in Foot Health Status Questionnaire pain domain | During baseline and at follow-ups after 4, 12, 26 and 52 weeks
  The Foot Health Status Questionnaire is a self-report questionnaire ranging from 0 (poor foot health) to 100 (optimum foot health) that assesses multiple dimensions of foot health and function. A validated Danish translation of the original questionnaire will be used.

SECONDARY OUTCOMES:
Change in Foot Health Status Questionnaire function domain | During baseline and at follow-ups after 4, 12, 26 and 52 weeks
  Ranging from 0 (poor foot health) to 100 (optimum foot health)
Change in Foot Health Status Questionnaire footwear domain | During baseline and at follow-ups after 4, 12, 26 and 52 weeks
  Ranging from 0 (poor foot health) to 100 (optimum foot health)
Change in Foot Health Status Questionnaire general foot health domain | During baseline and at follow-ups after 4, 12, 26 and 52 weeks
  Ranging from 0 (poor foot health) to 100 (optimum foot health)
Global Rating of Change | At follow-ups after 12, 26 and 52 weeks
  This will be used to measure the participants' self-reported recovery on a 7-point Likert scale ranging from "much improved" to "much worse". Participants are categorised as improved if they rate themselves as "much improved" or "improved" (category 6-7) and categorised as not improved if they rate themselves from "slightly improved" to "much worse" (category 1-5)
Time to Patient Acceptable Symptom State | From 0 to 52 weeks
  This will be used as a measure of when participants achieve a self-evaluated satisfactory result and feels no further treatment is needed; hence, it is not necessarily a measure of complete recovery
Change in Pain Self-Efficacy Questionnaire score | During baseline and at follow-ups after 4, 12, 26 and 52 weeks
  The Pain Self-Efficacy Questionnaire ranges from 0 (not at all confident) to 60 (completely confident) with lower scores indicating lower self-efficacy. A Danish translation of the original questionnaire, which has been validated in a Danish chronic pain population, will be used
Change in weekly light, moderate and vigorous physical activity level expressed as Metabolic Equivalents | Week 1 and Week 13 of the interventions
  Participants will be wearing a wrist-worn accelerometer ((ActiGraph wGT3X-BT (ActiGraph LLC, Pensacola, FL, USA)) during the first three weeks after baseline and again during the first three weeks after the 12-week follow-up.
Change in self-reported health state as measured by the EQ-5D-5L | During baseline and at follow-ups after 4, 12, 26 and 52 weeks

OTHER OUTCOMES:
Sick leave | During baseline and at follow-ups after 4, 12, 26 and 52 weeks
  Participants are asked how many days of sick leave they have had during the past 4 weeks due to their condition
Condition-related expenses | During baseline and at follow-ups after 4, 12, 26 and 52 weeks
  Participants are asked which expenses and the size they have had during the past 4 weeks due to their condition

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Rathleff, PhD, Study Chair — Aalborg University
Locations (1):
- Department of occupational therapy and physiotherapy, Aalborg University Hospital, Hobrovej 18-22, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Riel H, Vicenzino B, Olesen JL, Bach Jensen M, Ehlers LH, Rathleff MS. Does a corticosteroid injection plus exercise or exercise alone add to the effect of patient advice and a heel cup for patients with plantar fasciopathy? A randomised clinical trial. Br J Sports Med. 2023 Sep;57(18):1180-1186. doi: 10.1136/bjsports-2023-106948. Epub 2023 Jul 6. PMID 37414460
- [Derived] Riel H, Vicenzino B, Olesen JL, Jensen MB, Ehlers LH, Rathleff MS. Corticosteroid injection plus exercise versus exercise, beyond advice and a heel cup for patients with plantar fasciopathy: protocol for a randomised clinical superiority trial (the FIX-Heel trial). Trials. 2020 Jan 2;21(1):5. doi: 10.1186/s13063-019-3977-0. PMID 31898517